CLINICAL TRIAL: NCT03663140
Title: Neurogenic Inflammatory Response in Peri-implant and Periodontal Diseases Assessed by Biochemical Analysis of the Neuropeptides in Gingival Crevicular Fluid.
Brief Title: Neurogenic Inflammation in Peri-implant and Periodontal Diseases
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, muge lutfioglu, assoc. prof.dr, Ondokuz Mayıs University
Other Study IDs: OMU KAEK 2011/752
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Neurogenic Inflammation; Periimplant Diseases; Periodontal Diseases; Gingival Crevicular Fluid; Periimplant Sulcular Fluid
MeSH Terms: conditions — Neurogenic Inflammation; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — gingival crevicular fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1-Health periodontal: This group created by individuals with healthy periodontal tissues. Periodontal status/peri-implant was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  Interventions: Diagnostic Test: gingival crevicular fluid (GCF) and peri-implant sulcular fluid(PISF) collection
- Group 2- Healthy peri-implant: This group created by individuals with healthy peri-implant tissues. Periodontal status/peri-implant was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  Interventions: Diagnostic Test: gingival crevicular fluid (GCF) and peri-implant sulcular fluid(PISF) collection
- group 3- Gingivitis: This group created by individuals with gingivitis. Periodontal/peri-implant status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  Interventions: Diagnostic Test: gingival crevicular fluid (GCF) and peri-implant sulcular fluid(PISF) collection
- Group 4-Peri-implant Mucositis: This group created by individuals with peri-implant mucositis. Periodontal/peri-implant status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  Interventions: Diagnostic Test: gingival crevicular fluid (GCF) and peri-implant sulcular fluid(PISF) collection
- Group 5-Periodontitis: This group created by individuals with periodontitis. Periodontal/peri-implant status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  Interventions: Diagnostic Test: gingival crevicular fluid (GCF) and peri-implant sulcular fluid(PISF) collection
- Group 6-Periimplantitis: This group created by individuals with peri-implantitis. Periodontal/peri-implant status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  Interventions: Diagnostic Test: gingival crevicular fluid (GCF) and peri-implant sulcular fluid(PISF) collection

INTERVENTIONS:
Diagnostic Test: gingival crevicular fluid (GCF) and peri-implant sulcular fluid(PISF) collection — GCF/PISF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva.

SUMMARY:
Regulatory effects of some neuropeptides substance-P (SP), neurokinin-A (NKA), calcitonin gene-linked peptide (CGRP) and neuropeptide-Y (NPY) )on inflammatory responses in periodontal disease has been described; however, the impact of neuropeptide levels are not clearly defined in healthy and diseased peri-implant tissues.ın order to evaluate the situation, thirty-nine implants that have been loaded over the past 12 months and their symmetrically matching teeth were evaluated using a split-mouth study design. Clinical periodontal examinations included the Silness-Löe plaque index, Löe-Silness gingival index, bleeding on probing, probing pocket depth and clinical attachment level parameters were determined. Gingival crevicular fluid (GCF)/Periimplant sulcular fluid (PISF) samples were collected, and the levels of the neuropeptides were determined by enzyme-linked immunosorbent assay. Correlations between GCF/PISF neuropeptide levels and the clinical examination parameters were evaluated in the peri-implant/periodontal soft tissues.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria for patient selection were as follows:

* Compliance with systematic maintenance care;
* Adult, non-smoker, systemically healthy
* Not using any medicament for the last 6 months ;
* Partially dentated patient treated with implant-supported metal ceramic full crowns and/or fixed partial dentures
* As the study was split-mouth designed, in each individual at least one implant and one matching tooth in the same mouth symmetrically representing the same tooth group (premolars/molars);
* A single type of metal ceramic implant restoration that is functional for at least 1 year; and a matching tooth with no dental or endodontic restorations.

Exclusion Criteria:

* Medical history of cancer, rheumatoid arthritis, diabetes mellitus, or cardiovascular disease and any other systemic disease affecting lipid metabolism (i.e. impaired glucose tolerance, metabolic syndrome);
* Compromised immune system;
* Pregnancy, menopause, or lactation;
* Ongoing drug therapy that might affect the clinical characteristics of periodontitis and lipid metabolism;
* Dental treatment during the 6 months prior to data collection.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty-nine male, systemically healthy adult individuals (35-55 years old) and 39 dental implants were recruited for the present study. The same implant system was utilized for the treatments and the clinical treatment procedures were completed by the same two clinicians at the Ondokuz Mayis University Dental Faculty between 2011 and 2013.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-09-15 (Actual); Study Completion 2013-12-30 (Actual)

PRIMARY OUTCOMES:
Gingival crevicular fluid/peri-implant sulcular fluid Level of Substance-P | 8-10 am on the day following periodontal status assessment.
  Substance-P (SP) is a neuropeptide of the tachykinin family and marker of neurogenic inflammation.
Gingival crevicular fluid/peri-implant sulcular fluid Level of neurokinin-A | 8-10 am on the day following periodontal status assessment.
  Neurokinin-A is a neuropeptide of the tachykinin family and marker of neurogenic inflammation.
Gingival crevicular fluid/peri-implant sulcular fluid Level of Calcitonin gene-related peptide | 8-10 am on the day following periodontal status assessment.
  Calcitonin gene-related peptide (CGRP), another neuropeptide derived from peptidergic nerves and a marker of neurogenic inflammation.